CLINICAL TRIAL: NCT04455074
Title: French Validation Study of a New Scale for Neuropsychiatric Fluctuations in Parkinson Disease
Brief Title: Validation of the Neuropsychiatric Fluctuations Scale (EFN-VALID))
Acronym: EFN-VALID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC20.116; 2020-A00862-37 (Other: ID RCB)
Record Dates: First submitted 2020-04-23; First posted 2020-07-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease; Fluctuating Mood Symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD patients with motor fluctuations (Experimental): FN scale is an autoquestionnaire consisting of 20 questions, to be answered in On-med and OFF-med condition
  Interventions: Other: FN scale auto-questionnaire

INTERVENTIONS:
Other: FN scale auto-questionnaire — Patients will be asked to fill in the NF scale questionnaire together with other tests and rating scales, during a routine L-Dopa test, in 2 conditions: OFF-med and ON-med.

SUMMARY:
Neuropsychiatric fluctuations (NF) are among the most disabling non motor fluctuations in Parkinson disease (PD). The investigators developed the NF-scale for acute assessment of non-motor neuropsychiatric fluctuations between the off- and on-medication conditions in PD. The main goal of this project is to validate the NF-scale in french language in a multicenter approach.

DETAILED DESCRIPTION:
Anxiety, sadness, lack of energy and motivation, fatigue and pain are common during the off-medication condition, whereas euphoria, well-being, impulse control disorders, behavioral addictions, mania, and psychosis might occur during the on-medication condition. Early diagnosis of NpsyF is crucial for their holistic management. Unfortunately, NpsyF are often under-recognized by patients or misdiagnosed by physicians due to the lack of specific assessment tools. The NFS is composed of 20 items among which ten measure the "ON neuropsychological state" and ten, the "OFF neuropsychological state". It provides two sub-scores (one ON and one OFF) with a maximal total score of 30.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* presence of motor fluctuations, requiring a levodopa test
* french native speaker

Exclusion Criteria:

* Dementia (MoCa < 24)
* Parkinson syndrome other than idiopathic PD
* people excluded according to french law (including pregnant women or nursing mothers, ...)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
validation of FN scale: realiability | 2 months
  EFN score
validation of FN scale: internal consistency | 4 hours
  EFN score
validation of FN scale: measurement error | 2 months
  test-retest
validation of FN scale: structural validity | 4 hours
  EFN score
validation of FN scale: responsiveness | 4 hours
validation of FN scale: acceptability | 4 hours
  EFN score

SECONDARY OUTCOMES:
correlation of EFN scores with socio-clinical characteristics 1 | 4 hours
  MDS-UPDRS
correlation of EFN scores with socio-clinical characteristics 2 | 4 hours
  Severity of PD (Clinical Impression of Severity Index for PD - CISI-PD)
correlation of EFN scores with socio-clinical characteristics 3 | 4 hours
  stage of PD (Hoehn & Yahr stage)
correlation of EFN scores with socio-clinical characteristics (4) | 4 hours
  cognitif state (Montreal cognitive assessment - MoCA test)
correlation of EFN scores with socio-clinical characteristics (5) | 4 hours
  Impulsive-Compulsive Disorders (QUIP-RS)
correlation of EFN scores with socio-clinical characteristics (6) | 4 hours
  Dopamine-dependant behavior (ACDD)
correlation of EFN scores with socio-clinical characteristics (7) | 4 hours
  Wearing off (QUICK questionnaire)
correlation of EFN scores with socio-clinical characteristics (8) | 4 hours
  Depression (Beck depression inventory BDI-II)
correlation of EFN scores with socio-clinical characteristics (9) | 4 hours
  Evalulation of impulsive behavior (UPSS)

CONTACTS AND LOCATIONS:
Overall Officials: Elena MORO, MD PhD, Principal Investigator — University Hospital, Grenoble
Locations (6):
- France (6):
  - CHU Amiens, Amiens
  - CHU de Bordeaux-Hôpital Pellegrin, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - University hospital grenoble, Grenoble
  - Hospices Civils Lyon (HCL), Lyon
  - CHRU Strasbourg, Strasbourg

REFERENCES:
- [Result] Schmitt E, Bouvard M, Anheim M, Guehl D, Klinger H, Laurencin C, Marques A, Meissner WG, Thobois S, Thomas J, Tir M, Debu B, Moro E; NFS-VALID Study. Neuropsychiatric fluctuations in Parkinson's disease: A French multicenter study of the NFS psychometric properties. Parkinsonism Relat Disord. 2025 Sep;138:107954. doi: 10.1016/j.parkreldis.2025.107954. Epub 2025 Jul 11. PMID 40683099